CLINICAL TRIAL: NCT04386798
Title: Determination of Stress and Anxiety Levels of Mothers Lying in the Newborn Intensive Care Unit During Coronavirus Disease Pandemic Period
Brief Title: Stress and Anxiety Levels of Mothers Lying in the Baby Newborn Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, DILEK SAYIK, Nurse, Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DSAYIK1
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Newborn; Anxiety
Keywords: newborn intensive care; mother's anxiety; coronavirus pandemic
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- survey application to mothers (Other): In the neonatal intensive care, the information form, postpartum specific anxiety scale, and neonatal intensive care unit parent-father stress scale will be filled in for the mothers who have a baby.
  Interventions: Other: survey work

INTERVENTIONS:
Other: survey work — Bebeği Yenidoğan Yoğun Bakım Ünitesinde Yatan Annelerin Stres ve Anksiyete Düzeyleri anket yöntemi ile ölçülecektir.

SUMMARY:
Although coronaviruses (CoV) cause mild infections in the community, such as colds, they can also cause more severe infections. There are many subspecies of coronaviruses that can pass from animals to humans and can be transmitted between humans. One of these subspecies is COVID-19 (severe acute respiratory syndrome coronavirus 2), SARS-CoV-2, and has made a worldwide pandemic from the beginning of 2020. In this process, going out of the house, going to the hospital and being in the hospital brings with it the anxiety to get sick. In the period when the feeling of motherhood begins at the end of birth, the hospitalization of the baby for any reason and the separation of the mother and the baby can be an additional source of stress. This study was planned to determine the anxiety and anxiety levels of mothers who had a baby in the NICU during Coronavirus disease pandemic and the factors affecting them.

DETAILED DESCRIPTION:
Although coronaviruses (CoV) cause mild infections in the community, such as colds, they can also cause more severe infections. There are many subspecies of coronaviruses that can pass from animals to humans and can be transmitted between humans. One of these subspecies is COVID-19 (severe acute respiratory syndrome coronavirus 2), or SARS-CoV-2, and has made a worldwide pandemic from the beginning of 2020. Many countries are taking measures to protect everyone, including those in the risk group, to prevent disease in large groups and balance hospital bed capacities against the COVID-19 pandemic. Among these measures; There is an incentive for public health practices such as contact isolation, quarantine, frequent hand washing, not going out of the house unless needed, and social distance. In the investigator's country, preventive and therapeutic measures (such as quarantine, social distance) are taken against the COVID-19 pandemic and the public is constantly informed in this context. In this process, going out of the house, going to the hospital and being in the hospital brings with it the anxiety to get sick. Despite all these, there are compulsory situations requiring people to be in the hospital during the pandemic period. One of them is to give birth and then the baby stays in the hospital due to the need for intensive care.

Although it is a pleasant feeling for women who have just given birth to feel the feeling of motherhood, to embrace the baby, to attach it to the baby, adapting to the new situation with the accompanying responsibilities can force the mother psychologically In the period when the feeling of motherhood begins, the hospitalization of the baby for any reason and the separation of the mother and the baby may be an additional source of stress. The fact that this process is experienced during the pandemic period can increase the anxiety and stress in the mother much more. It is important for nurses to determine the needs of mothers whose babies are in the neonatal intensive care unit (NICU) during their pandemic, in order to reduce their anxiety and anxiety by applying appropriate nursing approach. This study was planned to determine the anxiety and anxiety levels of mothers who had a baby in the NICU during Coronavirus disease pandemic and the factors affecting them.

ELIGIBILITY:
Inclusion Criteria:

* Mothers whose babies are lying in YYBÜ,
* Agree to participate in the study,
* without communication problems (who can speak Turkish ... etc.)
* Mothers who can read and write

Exclusion Criteria:

* Does not agree to participate in the research,
* readable and illiterate
* mothers with communication problems (who do not speak Turkish, etc.)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2020-07-25 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2021-12-25 (Actual)

PRIMARY OUTCOMES:
Mothers' anxiety rate | 30 days
  During Coronavirus disease pandemic, anxiety rates of mothers lying on their babies in their NICUs were correlated with sociodemographic features.

CONTACTS AND LOCATIONS:
Overall Officials: DILEK SAYIK, expert nurse, Principal Investigator — Eskisehir City Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Eskisehir City Hospital, Odunpazari, Eskişehir
  - Eskisehir City Hospital, Eskişehir

IPD SHARING:
Plan to Share IPD: Yes
When the study is completed and published in the journal, it will be shared
Supporting Information: Study Protocol
Time Frame: When the study is completed and published in the journal, it will be shared

REFERENCES:
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Bedford J, Enria D, Giesecke J, Heymann DL, Ihekweazu C, Kobinger G, Lane HC, Memish Z, Oh MD, Sall AA, Schuchat A, Ungchusak K, Wieler LH; WHO Strategic and Technical Advisory Group for Infectious Hazards. COVID-19: towards controlling of a pandemic. Lancet. 2020 Mar 28;395(10229):1015-1018. doi: 10.1016/S0140-6736(20)30673-5. Epub 2020 Mar 17. No abstract available. PMID 32197103
- [Background] T.C. Sağlık Bakanlığı COVID-19 (SARS-CoV-2 Enfeksiyonu) Rehberi Bilim Kurulu Çalışması 14.04.2020, https://covid19bilgi.saglik.gov.tr/depo/rehberler/COVID-19_Rehberi.pdf.
- [Background] Hu D, Kong Y, Li W, Han Q, Zhang X, Zhu LX, Wan SW, Liu Z, Shen Q, Yang J, He HG, Zhu J. Frontline nurses' burnout, anxiety, depression, and fear statuses and their associated factors during the COVID-19 outbreak in Wuhan, China: A large-scale cross-sectional study. EClinicalMedicine. 2020 Jun 27;24:100424. doi: 10.1016/j.eclinm.2020.100424. eCollection 2020 Jul. PMID 32766539
- [Background] Ovalı, F. (2020). Yenidoğanlarda COVID-19 Enfeksiyonları. Anadolu Kliniği Tıp Bilimleri Dergisi, 25(1), 23-45
- [Background] Turan, T., & Başbakkal, Z. (2006). Yenidoğan yoğun bakım ünitesi anne-baba stres ölçeğinin geçerlilik ve güvenilirlik çalışması. Hacettepe Üniversitesi Hemşirelik Fakültesi Dergisi, 13(2), 32-42.